CLINICAL TRIAL: NCT04516213
Title: An Open-label, Single-arm Study to Evaluate the Tolerance and Safety of a Peptide-based Enteral Formula with Partially Hydrolyzed Guar Gum (PHGG) in the Nutritional Management of Tube-fed Children Aged 1-4 Years.
Brief Title: Study to Evaluate the Tolerance and Safety of a Peptide-based Enteral Formula with Partially Hydrolyzed Guar Gum (PHGG)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19.02.CLI
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Enteral formula tube feeding (Experimental): Enterally fed children, ages 1-4, with established enteral feeding access
  Interventions: Other: Enteral Formula With (PHGG)

INTERVENTIONS:
Other: Enteral Formula With (PHGG) — Pediatric subjects will be fed a Peptide-based Enteral Formula With Partially Hydrolyzed Guar Gum (PHGG)

SUMMARY:
This is a Multicenter, Open-label, Single-arm study evaluating the Tolerance and Safety of a Peptide-based Enteral Formula with Partially Hydrolyzed Guar Gum (PHGG) in the Nutritional Management of Tube-fed Children Aged 1-4 Years over a 7 day period.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent from subject and/or subject's parents or legally authorized representatives (LAR).
* Male or female, 12 to 48 months of age, inclusive.
* Subjects requiring enteral feeding for > 7 days (in hospital, long-term care facility or at home).
* Subjects receiving enteral tube-feeding (nasogastric feeding tube or percutaneous endoscopic gastrostomy [PEG] tube) to provide 90% or more of their nutritional needs at the time of study entry.
* Subject is clinically stable (i.e. absence of any significant gastrointestinal symptoms during the past 7 days), in the opinion of the investigator.

Exclusion Criteria:

* Subjects receiving partial or total parenteral nutrition (e.g. for short bowel syndrome and other causes of intestinal failure).
* Subjects with ongoing or intermittent significant gastrointestinal symptoms during the 7 days before enrollment.
* Oncology patients recovering from chemotherapy or radiotherapy for hematological malignancies or solid tumors (last treatment within 3 months of enrollment).
* Congenital immunodeficiency syndromes (SCID etc).
* Cystic fibrosis and other causes of fat malabsorption (lymphatic malformations/lymphangiectasis).
* Subjects with any clinically significant condition (e.g. severe malnutrition, congenital heart disease, etc) that, in the investigator's opinion, would preclude inclusion in the study.
* Subjects at risk for poor compliance to the study protocol in the investigator's opinion.
* Currently participating in another conflicting trial or participated in an investigational trial within 30 days of enrollment.
* Known hypersensitivity to PHGG or to any other ingredients in the investigational product.

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
GI Intolerance | 7 Days
  Occurrence of gastrointestinal intolerance (yes/no)

SECONDARY OUTCOMES:
Adverse Events | 7 Days
  Frequency and nature of adverse events
Energy Requirements Met | 7 Days
  The daily percentage of energy requirements
Change in Weight | 7 Days
  The change in weight over a 7-day period

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Minor, MMS, PA-C, Principal Investigator — Children's Center for GI and Nutrition
Locations (5):
- United States (5):
  - Children's Center for GI and Nutrition, Hollywood, Florida
  - The University of Chicago Medicine, Chicago, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - The Children's Mercy Hospital, Kansas City, Missouri
  - University of Utah Health Care - Huntsman Cancer Institute (HCI), Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Minor G, Sentongo T, Heine RG, Zemrani B. Tolerability and safety of a semi-elemental enteral formula with partially hydrolyzed guar gum (PHGG) in tube-fed children aged 1-4 years: An open-label, single-arm study. Clin Nutr ESPEN. 2023 Jun;55:392-399. doi: 10.1016/j.clnesp.2023.04.004. Epub 2023 Apr 21. PMID 37202073